CLINICAL TRIAL: NCT03196401
Title: A Pilot Study to Evaluate for the Abscopal Effect of Durvalumab (Anti-PD-L1) in Combination With Definitive Radiation Therapy in Solitary Bone Plasmacytoma With Limited Clonal Bone Marrow Plasmacytosis
Brief Title: A Study of Durvalumab (Anti-PDL1) Plus Radiation Therapy for the Treatment of Solitary Bone Plasmacytoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA recommendation
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-269
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Solitary Bone Plasmacytoma
Keywords: Durvalumb; Radiation Therapy; Clonal Bone Marrow Plasmacytosis; MEDI4736; 17-269
MeSH Terms: interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This is an open-label, single center, single-arm pilot study of checkpoint blockade therapy (anti-PD-L1) plus radiation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab Plus Radiation Therapy (Experimental): Durvalumab (1500mg administered intravenously every 28 days), concurrently with definitive radiation therapy to the solitary bone plasmacytoma to start within 14 days of the first dose of durvalumab.
  Interventions: Drug: Durvalumab; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Durvalumab — durvalumab 1500mg administered intravenously every 28 days, for a total of six doses
  Other Names: (MEDI4736)
Radiation: Radiation therapy — concurrent definitive radiation therapy to the bone plasmacytoma initiated within two weeks of starting

SUMMARY:
This study is being done to evaluate whether the combination of immune therapy and radiation therapy to plasmacytoma that can stimulate the immune system to attack and eliminate the abnormal cells in the bone marrow and perhaps delay or prevent the cancer from worsening. This study will evaluate whether the immune system responds to the combination of radiation with immunotherapy. It is possible that that the combination of immune therapy and radiation may not make any difference in whether or not the patient will develop multiple myeloma in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed plasmacytoma amenable for biopsy
* Detectable clonal bone marrow plasma cells by multicolor flow cytometry and less than 10% clonal plasma cells in a bone marrow biopsy by immunohistochemistry, morphology, or flow cytometry.
* Clinically safe to delay radiation for at least 2 weeks.
* ECOG performance status of 0-1.
* Anticipated lifespan greater than 3 month.
* Adequate organ function, as defined below:

  * Total bilirubin within normal ranges unless associated with hepatobiliary metastases or Gilbert syndrome, then total bilirubin ≤ 2 x ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
  * Creatinine ≤ 2.0 mg/dL
* Able and willing to give valid written informed consent.

Exclusion Criteria:

* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis, Crohn's disease], diverticulitis with the exception of a prior episode that has resolved or diverticulosis, celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener's syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis, uveitis; etc) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion: subjects with vitiligo or alopecia; subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement; or subjects with psoriasis not requiring systemic treatment.
* Current or prior use of immunosuppressive medication within 14 days prior to first dose of durvalumab. The following are exceptions to this criterion: intranasal, inhaled, topical or local steroid injections (eg. intra-articular injection); steroids as premedication for hypersensitivity reactions; systemic corticosteroid at physiologic doses not to exceed 10mg/day of prednisone or equivalent.
* Known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or evidence of active hepatitis B virus (HBV).
* History of hypersensitivity to durvalumab or any excipient
* History of hypersensitivity to the combination or comparator agent (If applicable) Receipt of live attenuated vaccination within 30 days prior the first dose of durvalumab.
* Female subjects who are pregnant, breast-feeding or female patients of reproductive potential who are not employing an effective method of birth control from starting dose of durvalumab (Cycle 1 Day 1), including dosing interruptions through 90 days after receipt of the last dose of durvalumab. Refrain from egg cell donation while taking durvalumab and for at least 90 days after the last dose of durvalumab.
* Male subjects who are not employing an effective method of birth control from starting dose of durvalumab (Cycle 1 Day 1), including dosing interruptions through 90 days after receipt of the last dose of durvalumab. Refrain from sperm donation while taking durvalumab and for at least 90 days after the last dose of durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Response assessment | up to 36 months from start of cycle 1
  Disease assessments are made according to IMWG criteria including criteria for minimal residual disease

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lesokhin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm